CLINICAL TRIAL: NCT00325884
Title: Long-term Outcomes of Patients After Coronary Bifurcation Stenting
Status: Completed | Type: Observational
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Scott Kinlay, Director, Cardiac Catheterization Laboratory, VA Boston Healthcare System
Other Study IDs: VABHS-IRB-1934
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Death; Myocardial Infarction
Keywords: coronary artery disease; bifurcation lesions; percutaneous interventions; stenting; outcomes; death; myocardial infarction
MeSH Terms: conditions — Coronary Artery Disease; Death; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the long-term clinical outcomes after stenting bifurcation coronary artery lesions, and to determine whether simple or more complex techniques are associated with a better clinical outcome. We will also assess the risk factors associated with poorer clinical outcomes

DETAILED DESCRIPTION:
Coronary artery disease affecting the branch points of coronary arteries (bifurcation lesions) has a higher rate of restenosis after angioplasty than disease in regions not involving branch points. Post-procedural angiographic outcomes and in-hospital outcomes have been documented for a variety of techniques, but none have examined the long-term clinical outcomes.

Long-term clinical outcomes are important from the patients point of view and also determine the use of resources. Knowledge of the long-term outcomes from the various techniques used to treat bifurcation lesions would be important in determining guidelines for the treatment of bifurcation lesions. If simple techniques offer similar or better outcomes than more complex strategies, then this would justify simpler techniques such as main vessel stenting that would use less resources, expose the patient to less radiation, and contrast related to prolonged angioplasty procedures.

Comparisons: We will compare the long-term outcomes of simple versus complex stent techniques, and determine other risk factors for long-term outcome

ELIGIBILITY:
Inclusion Criteria:

* de novo coronary artery lesion in a main branch with at least a 50% stenosis
* lesions involve the ostium of a side branch artery
* main branch and side branch with reference diameters of at least 2mm
* at least one stent used to treat the lesion

Exclusion Criteria:

* restenosis lesions
* reference side branch artery less than 2mm diameter
* multiple bifurcation lesions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient receiving drug eluting or bare metal coronary stents for coronary bifurcation lesions
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2001-08; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kinlay, MBBS, PhD, Principal Investigator — VA Boston Healthcare System
Locations (1):
- VA Boston Healthcare System, West Roxbury, Massachusetts, United States

REFERENCES:
- [Result] Zamani P, Kinlay S. Relationship of side-branch intervention and drug-eluting stents to long-term outcomes after coronary bifurcation stenting. J Am Coll Cardiol 2008; 51(suppl B): B50-B51
- [Result] Zamani P, Kinlay S. Long-term risk of clinical events from stenting side branches of coronary bifurcation lesions with drug-eluting and bare-metal stents: an observational meta-analysis. Catheter Cardiovasc Interv. 2011 Feb 1;77(2):202-12. doi: 10.1002/ccd.22750. PMID 20824754